CLINICAL TRIAL: NCT06841471
Title: Association Between Corneal Sensitivity, Nerve Morphology, Tear Film Homeostasis and Dry Eye Symptoms
Brief Title: Role of Corneal Nerves in Dry Eye Disease
Status: Recruiting | Type: Observational
Sponsor: Daniela Nosch (Other)
Responsible Party: Sponsor-Investigator, Daniela Nosch, Lecturer, University of Applied Sciences and Arts Northwestern Switzerland
Organization: University of Applied Sciences and Arts Northwestern Switzerland (Other)
Other Study IDs: 2024-01949; 2024-01949 (Registry Identifier: REGISTRY: Swissethics)
Record Dates: First submitted 2025-02-17; First posted 2025-02-24 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Dry Eye Disease (DED); Dry Eye; Dry Eye Sensation; Corneal Nerve
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: healthy adults
- DED group: Adults with Dry Eye following the TFOS DEWS II Diagnosis consensus

SUMMARY:
This study aims to determine whether corneal nerve function and morphology are affected by tear film instability and ocular surface homeostasis loss. Additionally, it seeks to investigate whether these factors vary based on the severity of dry eye symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Group with DED: Diagnosis of DED based on the TFOS DEWS II report
* Group without DED: No diagnosis of DED

Exclusion Criteria:

* Exclusion criteria:
* Systemic disease that may affect ocular health and innervation
* injury or history of operations on the anterior or posterior segment of the eye, which can affect the corneal structure and physiology
* regular application of systemic or ocular medication known to affect the tear film except from DED medications
* eye drops or makeup on the day of measurement.

Remarks:

Contact lens wearers are asked not to wear contact lenses for 1 week before the first appointment.

Participant with DED medications will be asked to use only conservative-free eye drops on the days of examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy adults as well as adult with dry eye disease
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Differences of corneal nerve function and morphology in relation with DED signs | within one week
  Correlation coefficient between corneal sensitivity and corneal nerve morphology, and variables related to tear film stability and corneal surface homeostasis.

SECONDARY OUTCOMES:
Differences of corneal nerve function and morphology in relation with DED symptoms | within one week
  Correlation coefficient between corneal sensitivity, corneal nerve morphology, and the severity of dry eye symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Optometrym FHNW, Olten, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Belmonte C, Nichols JJ, Cox SM, Brock JA, Begley CG, Bereiter DA, Dartt DA, Galor A, Hamrah P, Ivanusic JJ, Jacobs DS, McNamara NA, Rosenblatt MI, Stapleton F, Wolffsohn JS. TFOS DEWS II pain and sensation report. Ocul Surf. 2017 Jul;15(3):404-437. doi: 10.1016/j.jtos.2017.05.002. Epub 2017 Jul 20. PMID 28736339